CLINICAL TRIAL: NCT03447938
Title: The Minimally Invasive Coronary Surgery Compared to STernotomy Coronary Artery Bypass Grafting Randomized Controlled Trial
Brief Title: The Minimally Invasive Coronary Surgery Compared to STernotomy Coronary Artery Bypass Grafting Trial
Acronym: MIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: London Health Sciences Centre (Other); Heart Center Leipzig - University Hospital (Other); Fortis Escorts Heart Institute (Other); The Methodist Hospital Research Institute (Other); Carolinas Medical Center (Other); Gundersen Lutheran Health System (Other); Jilin Heart Hospital (Other); Far Eastern Memorial Hospital (Other); Medtronic (Industry); Apollo Hospitals Enterprise Limited (Other); Fresno Heart and Surgical Hospital (Unknown); Ichinomiya-Nishi Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180008
Record Dates: First submitted 2018-02-06; First posted 2018-02-27 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG with sternotomy (Active Comparator): Patients in this group will undergo coronary artery bypass grafting (CABG) in the usual way, through an incision in the middle of the chest, through the breastbone or sternum (conventional CABG).
  Interventions: Procedure: Conventional CABG
- Minimally-invasive CABG (Experimental): Patients in this group will undergo coronary artery bypass grafting (CABG) using a minimally-invasive approach (MICS CABG), through smaller incisions between the ribs.
  Interventions: Procedure: MICS CABG

INTERVENTIONS:
Procedure: MICS CABG — Coronary artery bypass grafting performed through small incisions between the ribs.
  Other Names: Minimally invasive coronary artery bypass grafting
  Arms: Minimally-invasive CABG
Procedure: Conventional CABG — Coronary artery bypass grafting performed through an incision through the sternum or breastbone.
  Other Names: coronary artery bypass grafting via sternotomy
  Arms: CABG with sternotomy

SUMMARY:
MICS CABG (Minimally invasive coronary surgery), where coronary artery bypass grafting (CABG) is completed through a small incision over the left chest, has evolved to become a safe and less invasive alternative to conventional sternotomy CABG. Several observational studies have suggested significantly shorter time to return to physical activity for MICS CABG patients compared to sternotomy CABG patients. A randomized study is warranted to validate these findings, provide higher level of evidence, and potentially lead to changes in practice. The MIST Trial is a multi-centre, prospective, open label, randomized control trial comparing quality of life and recovery in the early post-operative period, between patients undergoing MICS CABG versus patients undergoing sternotomy CABG. Patients referred for isolated CABG for multi-vessel coronary artery disease and deemed technically suitable for sternotomy CABG as well as for MICS CABG are considered for enrollment into the trial. Quality of life questionnaires (The SF-36, Seattle Angina Questionnaire and EQ-5D-5L) will be used to assess the quality of life and recovery in patients undergoing sternotomy CABG or MICS CABG at 1 month, 3 months, 6 months and 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Angiographically-confirmed multi-vessel coronary artery disease lesions with >=70% in at least 2 major epicardial vessels in 2 or more coronary artery territories (left anterior descending (LAD), circumflex (CX) and right coronary artery (RCA)) OR lesions >=50% in the left main (LM)
* Patients who, in the opinion of the investigator, are amenable for coronary surgery through either median sternotomy or minimally-invasive approach.
* Patients who are willing and able to comply with all follow-up study visits.

Exclusion Criteria:

* <18 years of age
* concomitant cardiac procedure with CABG (e.g. valve repair or replacement)
* Previous cardiac surgery, mediastinal irradiation, or significant trauma to the chest
* Contra-indications for MICS CABG, including: severe pectus excavatum; severe pulmonary disease; hemodynamically significant left subclavian stenosis; morbid obesity; severe left ventricular (LV) dysfunction; no adequate PDA or marginal branch target; absence of femoral pulse bilaterally.
* Contraindications for conventional CABG via sternotomy
* Concomitant life-threatening disease likely to limit life expectancy to <2 years
* Emergency CABG with hemodynamic compromise
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life - physical function | 4 weeks after surgery
  Comparison of the physical quality of life between the two groups four weeks after surgery using the physical function score of the 36-Item Short Form Health Survey (SF-36). The physical function score is a scale from 0 (poor physical function) to 100 (excellent physical function, with an average score of 50. It includes items that assess physical functioning, bodily pain, physical role functioning, vitality, and generaly health perceptions.

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) and Target Vessel Revascularization (TVR) | Through study completion, an average of 1 year after surgery.
  A composite endpoint of mortality, peri-operative myocardial infarction, non-peri-operative myocardial infarction, stroke, and new CABG or PCI associated with documented ischemia.
Number of bypass grafts | During coronary artery bypass surgery
  A comparison of the mean number of bypass grafts performed between the two groups
Percentage of arterial grafts | During coronary artery bypass surgery
  A comparison of the percentage of bypass grafts that are arterial between the groups
Intra-operative transfusion | During coronary artery bypass surgery
  A comparison of the number of transfusions during surgery between the groups
Post-operative transfusion | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  A comparison of the number of transfusions after surgery between the groups
Re-exploration for bleeding | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  The incidence of re-exploration for bleeding after surgery
Post-operative pain | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Measurement of patient's subjective assessment of their pain after surgery using a visual analog scale
Duration of intubation | Measured from the time of arrival in the Intensive Care Unit until the time patients are extubated, an average of 12 hours.
  Comparison of the average duration of intubation between groups
Length of ICU stay | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Comparison of the average number of days spent in Intensive Care Unit between groups
Length of hospital stay | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Comparison of the average number of days spent in hospital between groups
Atrial fibrillation | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Incidence of new-onset atrial fibrillation after cardiac surgery
Wound infection | During the first 2 months after surgery
  Incidence of wound infections in each group
Angina | 4 weeks after surgery
  Prevalence of anginal symptoms, as measured by the Seattle Angina Questionnaire. The SAQ includes scales that measure physical limitation, stability of angina, frequency of angina, satisfaction with treatment, and perception of disease, each of which is measured on a scale of 0 to 100 where higher scores indicate better function or health.
Quality of Life - mental function | 4 weeks after surgery
  Comparison of the mental quality of life between the two groups four weeks after surgery using the mental component score of the 36-Item Short Form Health Survey (SF-36). The mental function score is a scale from 0 (poor mental quality of life) to 100 (excellent mental quality of life), with an average score of 50. It includes items that assess vitality, general health perceptions, emotional role functioning, social role functioning, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (13):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Canada (2):
  - Division of Cardiac Surgery, University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
- Jilin Heart Hospital, Jilin, Jilin, China
- Germany (2):
  - Leipzig Heart Institute GmbH, Leipzig, Saxony
  - Robert-Bosch-Hospital, Stuttgart
- India (2):
  - Apollo Hospital, Bangalore, Bangalore, Karnataka
  - Manipal Hospitals, New Delhi, National Capital Territory of Delhi
- Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba, Japan
- National University Hospital (NUH) - Singapore, Singapore, Singapore
- Far-Eastern Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.